CLINICAL TRIAL: NCT03079869
Title: Transition to Ferric Citrate Among Hemodialysis and Peritoneal Dialysis Patients: A Phase 4 "Real World" Experience Study From Kaiser Permanente Southern California
Brief Title: Transition to Ferric Citrate Among Hemodialysis and Peritoneal Dialysis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Keryx Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: FeCitrate; 11035 (Other: Kaiser Permanente Southern California IRB)
Record Dates: First submitted 2017-03-01; First posted 2017-03-15 (Actual); Results first posted 2022-01-13 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Hyperphosphatemia
MeSH Terms: conditions — Hyperphosphatemia | interventions — ferric citrate

STUDY DESIGN:
Intervention Model Description: Prospective non-randomized cohort study of 6-9 months duration (active study period 6 months).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ferric Citrate (Other): Auryxia, 210 mg ferric iron tablets equivalent to 1 g of ferric citrate are supplied as 200 tablets in 400-cc high-density polyethylene bottles.
  Interventions: Drug: Ferric Citrate

INTERVENTIONS:
Drug: Ferric Citrate — One to two tablets of Ferric Citrate phosphorus binder administered by mouth before every meal to prevent dietary phosphorus absorption.
  Other Names: Auryxia

SUMMARY:
Transition to Ferric Citrate among Hemodialysis and Peritoneal Dialysis Patients: A Phase 4 "Real World" Experience Study from Kaiser Permanente Southern California

DETAILED DESCRIPTION:
PROTOCOL SUMMARY

Title: Transition to Ferric Citrate among Hemodialysis and Peritoneal Dialysis Patients: A Phase 4 "Real World" Experience Study from Kaiser Permanente Southern California

Short Title: FeCitrate

Protocol Number: KP FeCitrate

Study Phase: 4

Study Site(s): Los Angeles Kaiser Sunset Medical Center

Number of Subjects: 55

Study Arms: 1

Indication: Hyperphosphatemia in end stage renal disease

Primary Purpose: To evaluate the efficacy of ferric citrate for control of serum phosphorus levels and maintenance of adequate iron stores among dialysis-dependent patients before and after conversion from traditional phosphate binders in a "real world" environment

Overview of Study Design: Prospective non-randomized cohort study of 6-9 months duration (active study period 6 months).

Investigational Product Administration: One to two tablets of Ferric Citrate phosphorus binder administered by mouth before every meal to prevent dietary phosphorus absorption.

Study Endpoint: Mean serum phosphorus levels and rate of successful phosphorus control (<5.5mg/dl) 6 months before and after treatment with ferric citrate

Statistical Methods: Not powered to detect statistical significance

ELIGIBILITY:
Inclusion Criteria:

* Currently using 3 to 18 pills per day of calcium acetate, sevelamer, lanthanum, or calcium carbonate
* Mean serum phosphorus 4.0-<8.0 mg/dl for 6 months prior to enrollment
* No allergy to iron
* Mean corrected serum calcium > 8.0 mg/dl for 6 months prior to enrollment
* Mean PTH < 1000 pg/ml for 6 months prior to enrollment
* Mean ferritin < 1500 ng/ml and mean iron sat < 50% for 6 months prior to enrollment

Exclusion Criteria:

* History of gastrointestinal bleeding within past 6 months
* History of hospitalization for gastroparesis, bowel obstruction, or abdominal surgery within past 6 months
* Acute kidney injury equal to or less than 3 months before the initial screening date
* Active malignancy
* Functioning renal transplant
* Patients with iron overload syndrome (e.g., Hemochromatosis)
* History autoimmune disease, hemoglobinopathy, hemochromatosis, sickle cell disease
* Active or past history of calciphylaxis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-09-14 (Actual); Study Completion 2019-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Kumar, MD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Los Angeles Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study subjects who received either hemodialysis (HD) or peritoneal dialysis (PD) at Kaiser Permanente Southern California, Los Angeles Medical Center were eligible for recruitment.
Pre-assignment Details: No pre-assignment events. 55 subjects were enrolled.
Groups:
- Ferric Citrate - Hemodialysis; Ferric Citrate - Peritoneal Dialysis: Auryxia, 210 mg ferric iron tablets equivalent to 1 g of ferric citrate are supplied as 200 tablets in 400-cc high-density polyethylene bottles.
  Ferric Citrate: One to two tablets of Ferric Citrate phosphorus binder administered by mouth before every meal to prevent dietary phosphorus absorption.
Period: Overall Study
Arm/Group | Ferric Citrate - Hemodialysis | Ferric Citrate - Peritoneal Dialysis
Started | 28 | 27
Completed | 15 | 16
Not Completed | 13 | 11
Not completed — Adverse Event | 6 | 8
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Protocol withdrawal criteria-off drug > 2 weeks | 3 | 2

BASELINE CHARACTERISTICS:
Population: A total of 28 Hemodialysis (HD) patients were enrolled. Of these, 2 patients withdrew prior to receiving the study drug, 3 patients withdrew within the first 2 weeks due to adverse event, 2 patients withdrew themselves after 1 day. Only 1 of the 27 Peritoneal Dialysis (PD) patients enrolled in the study withdrew.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ferric Citrate - Hemodialysis | Ferric Citrate - Peritoneal Dialysis | Total
Number analyzed (Participants) | 21 | 26 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (13) | 57 (14) | 60 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 15 | 19 | 34
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 7 | 6 | 13
  African American | 6 | 3 | 9
  White | 7 | 14 | 21
  Unknown Race | 1 | 3 | 4
  Hispanic | 7 | 12 | 19
  Not Hispanic | 14 | 13 | 27
  Unknown Ethnicity | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 21 | 26 | 47
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.4 (4.7) | 27.8 (5.2) | 28.1 (4.9)
Smoking [Count of Participants; unit: Participants] | 10 | 6 | 16
Duration on Dialysis [Mean (Standard Deviation); unit: months] | 29 (32.1) | 41.4 (49.2) | 36.2 (42.5)
Diabetes [Count of Participants; unit: Participants] | 8 | 7 | 15
Cerebrovascular Disease [Count of Participants; unit: Participants] | 6 | 2 | 8
Congestive Heart Failure [Count of Participants; unit: Participants] | 5 | 4 | 9
Ischemic Heart Failure [Count of Participants; unit: Participants] | 2 | 2 | 4
Peripheral Vascular Disease [Count of Participants; unit: Participants] | 5 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Phosphorus Levels
Description: Serum phosphorus levels measured by mg/dL from the 6 months prior to enrollment were compared to serum phosphorus levels collected during the 6 months of ferric citrate use
Time Frame: 6 months
Population: The final analysis included 21 Hemodialysis and 26 Peritoneal Dialysis patients after exclusion of early dropouts. Wilcoxon signed rank test was used to compare pre-treatment and on-treatment
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Ferric Citrate - Hemodialysis | Ferric Citrate - Peritoneal Dialysis
Number analyzed (Participants) | 21 | 26
mg/dL
  Pre-treatment | 5.3 (1) | 5.6 (0.8)
  On-treatment | 5.4 (1.1) | 6 (1.8)

2. Secondary Outcome: Intravenous (IV) Iron
Description: The amount of intravenous (IV) iron in mg used per month by participants for 6 months before and 6 months on Ferric Citrate treatment.
Time Frame: 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/mo
Arm/Group | Ferric Citrate - Hemodialysis | Ferric Citrate - Peritoneal Dialysis
Number analyzed (Participants) | 21 | 26
mg/mo
  Pre-Treatment | 249.2 (215.6) | 21.2 (43.1)
  On-Treatment | 102 (137.5) | 11.6 (33.7)

3. Secondary Outcome: Erythropoiesis Stimulating Agents (ESA) Dose
Description: Mean Erythropoiesis Stimulating Agents (ESA) use from the 6 months prior to enrollment were compared to ESA use during the 6 months of ferric citrate use. The mean ESA dose units given to each participant per month was used in the analysis of this outcome.
Time Frame: 6 months
Population: The final analysis included 21 Hemodialysis and 26 Peritoneal Dialysis patients after exclusion of early dropouts. Wilcoxon signed rank test was used to compare pre-treatment and post-treatment.
Measure: Mean (Standard Deviation); unit: units/mo
Arm/Group | Ferric Citrate - Hemodialysis | Ferric Citrate - Peritoneal Dialysis
Number analyzed (Participants) | 21 | 26
units/mo
  Pre-Treatment | 28761.1 (41314.1) | 16724.4 (14042.3)
  Post-Treatment | 16525.8 (16917) | 16780.1 (13433.7)

4. Secondary Outcome: Median Pill Count
Description: median pill count of ferric citrate pills/day required to maintain phosphorus control
Time Frame: 6 months
Population: The final analysis included 21 Hemodialysis and 26 Peritoneal Dialysis patients after exclusion of early dropouts.
Measure: Median (Inter-Quartile Range); unit: tablets per day
Arm/Group | Ferric Citrate - Hemodialysis | Ferric Citrate - Peritoneal Dialysis
Number analyzed (Participants) | 21 | 26
tablets per day
  Phosphate binder pill count prior to Ferric Citrate use | 9.5 [6.8 to 13.8] | 6 [6.0 to 9.0]
  Phosphate binder pill count during Ferric Citrate use | 6.0 [4.5 to 9.0] | 4.5 [2.0 to 6.0]

ADVERSE EVENTS:
Time Frame: 7 months
Description: Adverse event (AE's) were included for all patient who received study drug for at least 1 day (n=54). After the baseline visit adverse events are collected on a weekly basis for the hemodialysis patients, and on a bi-monthly basis from the dialysis patients, and again 30days after the termination of the study.
Arm/Group | Ferric Citrate - Hemodialysis | Ferric Citrate - Peritoneal Dialysis
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 7/27 | 10/27
Other Adverse Events (participants affected / at risk) | 23/27 | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ferric Citrate - Hemodialysis (N=27) | Ferric Citrate - Peritoneal Dialysis (N=27)
Arteriovenous fistula (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Congestive heart failure exacerbation (Cardiac disorders) | 0 (0) | 1 (1)
gallstone pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal swelling (General disorders) | 0 (0) | 1 (1)
Peritonitis (General disorders) | 0 (0) | 1 (1)
Right foot infection (Infections and infestations) | 0 (0) | 1 (1)
Chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — non-cardiac
Chronic back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intertrochanteric fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Left foot pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Right hip osteoporotic Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Laparoscopic right nephrectomy (Renal and urinary disorders) | 1 (1) | 0 (0)
Placement of catheter for HD (Renal and urinary disorders) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Right sided pleuroperitoneal leak (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Left heel ulcers (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Critical limb ischemia (Vascular disorders) | 1 (1) | 0 (0)
Hemorrhagic cerebrovascular accident (Vascular disorders) | 0 (0) | 1 (1)
Peripheral vascular disease (Vascular disorders) | 1 (1) | 0 (0) — from diabetes mellitus type 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ferric Citrate - Hemodialysis (N=27) | Ferric Citrate - Peritoneal Dialysis (N=27)
Black stool (Gastrointestinal disorders) | 20 | 25
Diarrhea (Gastrointestinal disorders) | 10 | 10
Constipation (Gastrointestinal disorders) | 4 | 5
Bloating/Gas (Gastrointestinal disorders) | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Nausea, vomiting (Gastrointestinal disorders) | 1 | 4
Decreased appetite (Metabolism and nutrition disorders) | 0 | 3
Itching/rash (Skin and subcutaneous tissue disorders) | 2 | 4
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Urinary Tract Infection (Renal and urinary disorders) | 1 | 0
Abscess (Infections and infestations) | 0 | 1
Peritonitis (General disorders) | 0 | 1
Chest Pain/Palpitations (Cardiac disorders) | 0 | 1
Fatigue (General disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-05): https://cdn.clinicaltrials.gov/large-docs/69/NCT03079869/Prot_SAP_000.pdf